CLINICAL TRIAL: NCT05439616
Title: An 8-Week, Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Phase 3 Study of the Efficacy and Safety of Cariprazine in the Treatment of Pediatric Subjects (5 to 17 Years of Age) With Autism Spectrum Disorder
Brief Title: Study of Cariprazine Oral Capsules or Solution to Assess Adverse Events and Change in Irritability Due to Autism Spectrum Disorder (ASD) in Participants Aged 5-17 Years With ASD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M21-465
Record Dates: First submitted 2022-06-28; First posted 2022-06-30 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Cariprazine; VRAYLAR; AGN-241780
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — cariprazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cariprazine (Experimental): Participants will receive age-and weight dependent flexible doses of cariprazine once daily for 8-weeks.
  Interventions: Drug: Cariprazine
- Placebo (Placebo Comparator): Participants will receive placebo once daily for 8-weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cariprazine — Oral Capsules or Oral Solution
  Other Names: VRAYLAR; AGN-241780
  Arms: Cariprazine
Drug: Placebo — Oral capsules or Oral Solution
  Arms: Placebo

SUMMARY:
Autism spectrum disorder (ASD) consists of deficits in social, communication, and cognitive development, repetitive and stereotypic behaviors. Many ASD patients show notably high levels of irritability, including verbal and physical aggression, self injury, and/or property destruction. Autistic infants tend to avoid eye contact and show little interest in others. This study will assess how safe and effective cariprazine is in treating pediatric participants (5 to 17 years of age) with ASD. Adverse events and change in disease activity will be assessed.

Cariprazine is an investigational drug being developed for the treatment of irritability due to ASD. This study is double-blinded means that neither the participants nor the study doctors will know who will be given cariprazine and who will be given placebo (does not contain treatment drug). Study doctors put the participants in 1 of the 2 groups, called treatment arms. Each group receives a different treatment. There is a 1 in 2 chance that participants will be assigned to placebo. Approximately 152 participants diagnosed with ASD will be enrolled in approximately 40 sites globally.

Participants will receive oral capsules or oral solution of cariprazine or placebo once daily for 8-weeks and will undergo a 4-week safety follow-up period.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participants at the time of screening must have a Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnosis of ASD, confirmed by Kiddie Schedule for Affective Disorders and Schizophrenia-Present and Lifetime (K-SADS-PL) administered at screening (Visit 1) by a trained clinician.
* Participants must have an Aberrant Behavior Checklist, 2nd edition - Community Version - Irritability (ABC-I) subscale score ≥ 18 (Visits 1 and 2).
* Participants must have a Clinical Global Impressions - Severity - Irritability (CGI-S Irritability) score ≥ 4 at screening (Visits 1 and 2).

Exclusion Criteria:

* Participants with diagnosis of intellectual disability (Intelligence quotient < 25).
* No history of major depressive disorder, bipolar disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, brief psychotic disorder, or psychotic disorder due to another medical condition, as excluded by administration of Kiddie Schedule for Affective Disorders and Schizophrenia-Present and Lifetime (K-SADS-PL).
* History of ASD that is associated with Rett Disorder, Fragile-X Syndrome, or Childhood Disintegrative Disorder.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 161 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-10-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Aberrant Behavior Checklist, 2nd edition - Community Version - Irritability (ABC-I) Subscale Score | Baseline (Week 0) to Week 8
  The Aberrant Behavior Checklist (ABC) - Community version is a 58-item, caregiver-rated scale designed to measure inappropriate and maladaptive behavior of people with developmental disabilities (including intellectual disability and ASD). The ABC has 5 subscales (Irritability, Social Withdrawal, Stereotypic Behavior, Hyperactivity and Inappropriate Speech). The caregiver rates the child's behavior from 0=not at all a problem to 3= the problem is severe in degree. The range for Irritability is 0 to 45. Higher scores indicate greater severity.

SECONDARY OUTCOMES:
Percentage of Participants with responder status of "Very Much Improved" or "Much Improved" on the Clinical Global Impression- Change Irritability (CGI-C Irritability) Scale | Week 8
  The Clinical Global Impression - Change-Irritability (CGI-C Irritability) is a single-item rating scale that assesses change in the severity of a participant's irritability from the clinician's perspective. The CGI-C Irritability 7-point graded response scale (1 = "Very much improved," 2 = "Much improved," 3 = "Minimally improved," 4 = "No change," 5 = "Minimally worse," 6 = "Much worse," or 7 = "Very much worse").
Change from Baseline in Parent-Rated Anxiety Scale for Youth with Autism Spectrum Disorder (PRAS-ASD) Total Score | Baseline (Week 0) to Week 8
  PRAS-ASD is a 25-item caregiver-reported measure of anxiety in participants aged 3 to 17 with ASD. All items use a 4-point response scale: 0 = "None (not present);" 1 = "Mild (present sometimes, not a real problem);" 2 = "Moderate (often present and a problem);" 3 = "Severe (very frequent and a major problem)." Total score ranges from 0 to 75, with higher scores indicating greater severity of anxiety.
Change from Baseline in Caregiver Strain Questionnaire Short Form 7-Item (CGSQ SF-7) total score | Baseline (Week 0) to Week 8
  CGSQ SF-7 is a caregiver-reported 7-item measure of self-reported strain that focuses on the impact of caring for a child with emotional and behavioral problems. Responses are scored on a 5-point scale (1 = "Not at all," 2 = "A little;" 3 = "Somewhat;" 4 = "Quite a bit;" and 5 "Very much") with higher scores indicating greater caregiver strain.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (36):
- United States (34):
  - Advanced Research Center /ID# 245049, Anaheim, California
  - Sun Valley Research Center /ID# 243133, Imperial, California
  - CHOC Children's Hospital /ID# 245577, Orange, California
  - Pacific Clinical Research Management Group /ID# 243019, Upland, California
  - D&H Doral Research Center-Doral /ID# 255457, Doral, Florida
  - Sarkis Clinical Trials /ID# 242868, Gainesville, Florida
  - Advanced Research Institute of Miami /ID# 243179, Homestead, Florida
  - Sandhill Research LLC /ID# 245079, Lake Mary, Florida
  - Axcess Medical Research /ID# 244952, Loxahatchee Groves, Florida
  - G+C Research Group, LLC /ID# 252016, Miami, Florida
  - Medical Research Group of Central Florida /ID# 243170, Orange City, Florida
  - K2 Medical Research - Orlando - South Orlando Avenue /ID# 248694, Orlando, Florida
  - APG Research, LLC /ID# 243130, Orlando, Florida
  - Nona Pediatric Center /ID# 245078, Orlando, Florida
  - Asclepes Research Centers - Spring Hill /ID# 248682, Spring Hill, Florida
  - D&H Tamarac Research Center /ID# 250436, Tamarac, Florida
  - Atlanta Center for Medical Research /ID# 243124, Atlanta, Georgia
  - Atlanta Behavioral Research, LLC /ID# 243082, Dunwoody, Georgia
  - iResearch Savannah /ID# 254582, Savannah, Georgia
  - Alivation Research /ID# 242915, Lincoln, Nebraska
  - Dr. Hosneara, M.D. LLC /ID# 252129, Jackson Heights, New York
  - Richmond Behavioral Associates An Evolution Research Group Portfolio Company /ID# 259578, Staten Island, New York
  - New Dawn Psychiatric Services PLLC /ID# 243697, Kinston, North Carolina
  - Quest Therapeutics of Avon Lake /ID# 252013, Avon Lake, Ohio
  - Cincinnati Children's Hospital /ID# 243968, Cincinnati, Ohio
  - CincyScience /ID# 242993, West Chester, Ohio
  - BioBehavioral Research of Austin /ID# 255460, Austin, Texas
  - Relaro Medical Trials /ID# 243126, Dallas, Texas
  - Cedar Health Research /ID# 248683, Dallas, Texas
  - AIM Trials /ID# 243120, Plano, Texas
  - Family Psychiatry of The Woodlands /ID# 242867, The Woodlands, Texas
  - Advanced Research Institute /ID# 243098, Ogden, Utah
  - Northwest Clinical Research Center /ID# 243083, Bellevue, Washington
  - Core Clinical Research /ID# 243084, Everett, Washington
- Puerto Rico (2):
  - Dr. Samuel Sanchez PSC /ID# 245739, Caguas
  - GCM Medical Group PSC /ID# 245735, San Juan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M21-465